CLINICAL TRIAL: NCT06894680
Title: The Adaptation of a Stepped Care, Task-sharing Approach for Integrating Depression Care for Older People Living With HIV (PLHIV) Into HIV Treatment and Support Services in Ibadan, Nigeria.
Brief Title: Integrating Depression Care Into HIV Services for Older People With HIV Using a Stepped Care, Task-Sharing Approach.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Society of Tropical Medicine and Hygiene (Other)
Responsible Party: Principal Investigator, OLUFISAYO ELUGBADEBO, Dr, Royal Society of Tropical Medicine and Hygiene
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: SC-Depression-HIV-Ibadan-2025; NIhr24156 (Other Grant/Funding Number: NIHR)
Record Dates: First submitted 2025-03-18; First posted 2025-03-25 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Older Adults (50-90 Years); Depression
Keywords: Stepped-care approach; HIV and mental health; Older adults living with HIV(PLHIV); Depression care; Implementation research
MeSH Terms: conditions — Depression; Psychological Well-Being | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as Usual (Active Comparator): Participants in the Treatment as Usual arm will receive the routine care available for people living with HIV with depression at the health facility.
  Interventions: Other: Treatment as usual
- Intervention arm (Experimental): Step 1 at baseline PHQ-9 ≥10-14: Psychosocial intervention (PI) only for 6 weeks. PHQ-9 ≥15: supervising psychiatrist review + anti-depressants(sertraline) + PI for 6 weeks.
  At 6 weeks assessment, if PHQ-9 is ≥10; proceed to step 2. Others with PHQ<10: Continue bi-weekly PI to complete 3rd & 6th month assessment.
  Step 2
  1. PHQ-9 ≥10 (without previous antidepressant); supervising psychiatrist review + antidepressants + weekly PI for 6 weeks (to complete 3rd month assessment).
  2. PHQ-9 ≥10 (with previous antidepressant use); supervising psychiatrist to review medication + weekly PI for 6 weeks. At reassessment (3rd month assessment) if PHQ-9 ≥10; proceed to step 3.
  Others with PHQ<10 at 3rd month assessment: Continue bi-weekly follow-up and complete 6-month assessment.
  Step 3:
  PHQ-9 ≥10; supervising psychiatrist review every 6 weeks +antidepressant+ 2 PI per week At reassessment, participants with no improvement (PHQ-9 ≥10) ; refer to psychiatrist.
  Interventions: Other: Stepped care

INTERVENTIONS:
Other: Stepped care — It is a systematic, staged approach to delivering care based on the severity of a condition and the patient's response to treatment. In this model, less intensive interventions are provided first, and only those who do not improve progress to more intensive treatments.
  In clinical research, stepped-care is classified as an adaptive intervention, where treatment is adjusted based on pre-specified criteria, making it patient-centered and resource-efficient.
  Arms: Intervention arm
Other: Treatment as usual — Clients that are considered to be depressed are offered counselling by the Nurses who are the first point of contact. Depending on the severity of symptoms the client are then referred to the medical officer at the HIV clinic for assessment and offered counselling services by the counsellors. if symptoms are severe and considered to need specialist care the medical officer will refer to a specialist(psychiatrist) outside the HIV care facility.
  Arms: Treatment as Usual

SUMMARY:
Depression levels will be compared using PHQ-9 in the Treatment as Usual arm(TAU) VS intervention arm to see if the stepped care intervention is effective in treating depression. The main questions it aims to answer are:

* Needs assessment of stepped-care integration versus usual care for treating depression in older adults living with HIV?
* How effective will the stepped care task-sharing (SCT) model in reducing depressive symptoms and improving HIV treatment outcomes in older PLHIV in Nigeria? Participants who screen positive for depression PHQ-9 ≥10 will be randomized into 2 arms for treatment using a systemized ballot system: TAU arm and Intervention arm.

TAU arm will receive current treatment available for depression at the HIV center.

Intervention arm will receive the stepped-care intervention in stages based on their symptom severity.

Follow-up assessments at (6 weeks, 3months and 6 months) will be conducted by assessors who would be blinded to the different groups (TAU arm VS intervention arm).

DETAILED DESCRIPTION:
Depression is a common but often overlooked comorbidity among older adults living with HIV (PLHIV), particularly in low-resource settings. It negatively impacts health outcomes, adherence to antiretroviral therapy (ART), and overall quality of life. Despite its high prevalence, access to specialized mental health services remains limited due to workforce shortages and structural barriers within healthcare systems. A stepped-care task-sharing approach offers a potentially scalable solution by leveraging non-specialist healthcare workers to deliver evidence-based mental health interventions in a structured, stepwise manner. This study aims to evaluate the effectiveness of this approach in reducing depression among older PLHIV and assess its feasibility for broader implementation in Nigerian health facilities.

Study Objectives:

1. Effectiveness Assessment: To determine whether integrating a stepped-care task-sharing approach into routine HIV care is more effective in reducing depression symptoms compared to usual treatment among older PLHIV.
2. Implementation Feasibility: To identify facilitators and barriers to the successful adaptation and implementation of this intervention in local HIV facilities.
3. Patient Outcomes & Treatment Pathways: To evaluate the impact of the intervention on depression severity using the Patient Health Questionnaire-9 (PHQ-9) and examine how patients progress through different treatment steps based on symptom severity.

Study Design & Methodology:

This is a randomized controlled trial (RCT) comparing a stepped-care task-sharing intervention to usual care in older PLHIV with depressive symptoms.

* Inclusion criteria:

  o Older adults (≥50 years) living with HIV who screen positive for depression using PHQ-9.
* Randomization:

  o Participants will be randomly assigned to either the intervention arm (stepped-care intervention) or the control arm (treatment as usual).
* Intervention Model:

  * The intervention follows a stepped-care framework, where treatment intensity is adjusted based on depression severity at each stage.

Outcome Measures:

1. Primary Outcome

   o Reduction in depression severity as measured by PHQ-9 at 6 weeks, 3 months, and 6 months.
2. Secondary Outcomes

   * Acceptability of intervention.
   * Barriers and facilitators to implementation (qualitative analysis).
   * Changes in quality of life and HIV treatment adherence.

The RE-AIM (Reach, Effectiveness, Adoption, Implementation and Maintenance) framework will be used to evaluate effectiveness and implementation and will be measured using the following endpoints:

1. Identify barriers and facilitators in adapting a stepped care task-sharing model for depression care.

   End point: Identify barriers and facilitators in adapting a stepped care task-sharing model for depression care. Effectiveness is determined by comparing:

   Primary Outcome: Reduction in PHQ-9 scores (depression severity).

   Secondary Outcomes:

   Adherence to psychosocial intervention sessions and medication.

   Secondary objectives:
2. To compare the effectiveness of utilizing a stepped care task-sharing (SCT) model to usual treatment depression in older PLHIV in an HIV clinic in Nigeria.

Primary outcome: Rates of reduced depressive symptoms.

Secondary outcomes:

Assessing the rates of reduction in depressive symptoms from baseline to after intervention.

Significance of the Study This trial will provide evidence on the effectiveness and feasibility of integrating depression care within routine HIV services using a stepped-care, task-sharing model in Nigeria.

ELIGIBILITY:
Inclusion Criteria:

* Consenting individuals living with HIV
* People living with HIV who are 50 years and above (PLHIV aged ≥50 years)
* Those with a score of ≥10 on the 9-item patient-health questionnaire (PHQ-9).

Exclusion Criteria:

* • Older PLHIV will be assessed for the imminent risk of suicide and if there is an high risk, participant will be excluded.

  * Older PLHIV with severe cognitive impairment or diagnosed dementia that limits their ability to provide informed consent or complete study visits will be excluded.
  * Participants with comorbidities that can preclude the use of sertraline should be excluded.

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-24 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of a Stepped-Care Task-Sharing (SCT) Model in reducing depressive symptoms measured by PHQ-9. | Baseline PHQ-9 score (before intervention) Follow-up assessments at 6 weeks, 3 months, and 6 months
  This outcome will determine whether the Stepped care task-sharing approach provides greater symptom relief compared to usual treatment and supports its potential integration into routine HIV treatment and support service.

CONTACTS AND LOCATIONS:
Overall Officials: Olufisayo O Elugbadebo, MBBS, Msc, Principal Investigator — Department of Psychiatry, College of Medicine, University of Ibadan, Nigeria
Locations (1):
- Institute of Infectious Diseases, Ibadan, Oyo State, Nigeria

IPD SHARING:
Plan to Share IPD: No